CLINICAL TRIAL: NCT06249256
Title: An Exploratory Study on the Treatment of Advanced Solid Tumors by Secretory PD1 Nanoantibody Targeting Mesothelin Fast CAR T Cells
Brief Title: An Exploratory Study on the Treatment of Advanced Solid Tumors by Fast CAR T Cells
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZT2312-A-01
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fast CAR T cells (Experimental): The safety and efficacy of BZT2312 will be assessed in a standard 3+3 dose escalation approach. Three doses of CAR T cells will be evaluated in this study: 5×10^5 CAR+ T cells/kg, 1×10^6 CAR+ T cells/kg, and 5×10^6 CAR+ T cells/kg.
  Interventions: Biological: Fast CAR T cells

INTERVENTIONS:
Biological: Fast CAR T cells — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of Fast CAR T cells. During Fast CAR T cells production, subjects will receive cyclophosphamide and fludarabine for the purpose of lymphocytes depletion. After lymphodepletion, subjects will receive one dose treatment with Fast CAR T cells by intravenous (IV) injection.

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and tolerability of fast autologous mesothelin (MSLN)-targeted chimeric antigen receptor (MSLN-CAR) T cells secreting PD-1 nanobodies in patients with solid tumors.

DETAILED DESCRIPTION:
The main aim of this study is to determin the safety and efficacy of BZT2312 in patients with solid tumors. BZT2312 is an autologous mesothelin (MSLN)-targeted chimeric antigen receptor (MSLN-CAR) T cells secreting PD-1 nanobodies.

This study comprises of a screening phase(less than or equal to 28 days prior to apheresis) followed by apheresis(will occur upon enroiiment); Apheresis phase(less than or equal to 10 days prior to infusion ) followed by lymphodepletion. lymphodepletion phase (from day -5 to day -3) followed by infusion.Treatment Phase including infusion of BZT2312 on Day0 and then post-infusion assessments from Day1 to Day 28; and a Post-treatment Phase(Day 29 and up to end of the study). Efficacy will be explored to assessed and safety will be closely monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced solid tumors through histopathological diagnosis have a positive rate of ≥ 50% for mesothelin expression membrane in tumor tissue samples, PD-L1 positive expression, and sample sources within 2 years；
* Late stage malignant solid tumor patients who have failed standard treatment or are intolerant to such treatment and do not have a standard effective treatment plan；
* Greater than or equal to 18 years of age and less than or equal to 70 years of age on day of signing informed consent；
* Life expectancy >3 months；
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
* Satisfactory organ and bone marrow function as defined by the following:

  1. absolute neutrophil count must be greater than ≥ 1.5×109/L, lymphocyte count must be greater than ≥ 0.5×109/L, platelets must be greater than ≥ 90×109/L, hemoglobin must be greater than ≥ 90g/L without transfusion within 7 days or dependency on EPO;
  2. Total bilirubin must be less than or equal to two times (≤2.0x) the institutional normal upper limit; transaminases, serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST), must be less than or equal to 2.5 times (≤2.5x) the institutional normal upper limit (≤5x if there is hepatic metastasis);
  3. International normalized ratio (INR) or the PT is not greater than one and one half times (≤ 1.5) the upper limit of normal;
  4. Lung function: ≤ CTCAE grade 1 dyspnea and SaO2≥ 91%
  5. Cardiac function: cardiac ejection fraction (LVEF) must be greater than fifty percent (≥50%) by echocardiogram or MUGA one month before enrollment.
* Subjects must have measureable disease as defined by RECIST 1.1 criteria;
* Subjects sufficiently understand the trial and willingly sign the informed consent；
* Male and Female subjects agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) during the study and for at least 12 months following the last dose of the study cell infusion and until no CAR-T cells can be detected after two consecutive PCR tests.

Exclusion Criteria:

* Subjects who have undergone other anti-tumor treatments (including radiation therapy, chemotherapy, small molecule, biological or immunotherapy, and other study drugs) other than lymphocytes depletion allowed by the protocol within one month prior to CAR-T infusion;
* Prior therapy with any gene therapy (including CAR-T cell therapy) or any T cell therapy home and abroad;
* Pregnant or breastfeeding women;
* Positive serological reactions for HIV and syphilis; Hepatitis B surface antigen positive, hepatitis B core antibody positive, and hepatitis B virus DNA copy number higher than the detection limit and/or greater than or equal to 1000 copies/mL; Or Hepatitis C virus infected individuals;
* Any uncontrollable active infection, coagulation disorders, or any other major illness;
* Patients with autoimmune diseases, organ transplantation and other immune related diseases under treatment, or long-term use of immunosuppressive drugs such as glucocorticoids: a. Glucocorticoids: users cannot stop using CAR-T cells 72 hours before infusion; b. Immunosuppressants other than glucocorticoids cannot be stopped ≥ 4 weeks before enrollment;
* Patients who are allergic to BZT2312 components;
* History of severe cardiac or pulmonary disease, including hypertension that cannot be controlled by medication, and any of the conditions occurred within the past 6 months: congestive heart failure (New York Heart Association functional classification ≥3), cardiac angioplasty and stents, myocardial infarction, unstable angina, or other clinically significant heart disease;
* Detectable clinically relevant central nervous system (CNS) metastases and/or pathology such as epilepsy/seizure, brain Ischemia/ hemorrhage, dementia, cerebellar disease, or autoimmune disease affecting central nervous system
* Patients at high risk of causing bleeding or perforation;
* Patients who had undergone major surgical procedures or significant trauma within 4 weeks before apheresis, or who were expected to require major surgery during the study period;
* Patient has a known history of a hematologic malignancy, or of another malignant primary solid tumor concurrently, with the exception of :Patients with in situ cervical cancer or breast cancer with no evidence of disease for ≥ 3 years after curative treatments;Patients who underwent successful definitive resection of in situ cancer with no evidence of disease for ≥5 years;
* Other circumstances that were deemed by the investigator to be inappropriate for trial participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 28 days
  Safety

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days
  Tolerability
Objective response rate (ORR) | Month 12
  Clinical response will be assessed by RECIST 1.1
Progression-free survival (PFS) | Month 12
  PFS of patients receiving Fast CAR T cells
Overall survival (OS) | Month 12
  OS of patients receiving Fast CAR T cells
Peak Plasma Concentration (Cmax) | Month 12
  Pharmacokinetics (PK)
AUC | Month 12
  Pharmacokinetics (PK)
Pharmacodynamics (PD) | Day 28
  D of IL-2, IL-4, IL-6, IL-8, IL-10, IL-15, IFN-γ, TNF-α and MCP1 will be analysed after CAR T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jinxing Lou, Principal Investigator — Shanghai Mengchao Cancer Hospital
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No